CLINICAL TRIAL: NCT01164319
Title: Typing of the Atrial Fibrillation Recurrences in Early Postoperative Period After Pulmonary Veins Isolation Through Continous Subcutaneous Monitoring.
Brief Title: "UNMASKING Study" For Atrial Fibrillation Recurrences Typing in Early Postoperative Period
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AFERAWCLP-022; RU AF 002 (Other: State Research Institute of Circulation Pathology)
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Percutaneous continous monitoring; ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (no early recurrence) (Active Comparator): Patients without atrial fibrillation recurrences through the implantable cardiac monitors during the 3 months post-ablation period.
  Interventions: Procedure: Circumferential PVI and subcutaneous cardiac monitor implantation
- Group 2 (early AF recurrence) (Active Comparator): Patients with AF recurrences documented by the ICM during the 3 months post-ablation period.
  Interventions: Procedure: Circumferential PVI and subcutaneous cardiac monitor implantation
- Group 3 (early recurrence-no reablation) (Active Comparator): Patients with AF recurrences documented by the ICM during the 3 months post-ablation period from Group 2 would not receive reablation.
  Interventions: Procedure: Circumferential PVI and subcutaneous cardiac monitor implantation
- Group 4 (early recurrence-early reablation) (Active Comparator): Patients with AF recurrences documented by the ICM during the 3 months post-ablation period from Group 2 will receive early reablation based on data stored by implanted monitor.
  Interventions: Procedure: Circumferential PVI and subcutaneous cardiac monitor implantation

INTERVENTIONS:
Procedure: Circumferential PVI and subcutaneous cardiac monitor implantation — The left atrium (LA) and PVs were explored through a transeptal approach. Real-time 3D LA maps were reconstructed by using a nonfluoroscopic navigation system (CARTO, Biosense-Webster Inc.). The ipsilateral left and right PVs were encircled in one lesion line by circumferential PV isolation. Radiofrequency energy was delivered at 43°C, 35 W, 0.5 cm away from the PV ostia at the anterior wall, and was reduced to 43°C, 30 W, 1 cm away from the PV ostia at the posterior wall, with a saline irrigation speed of 17 mL/min. The endpoint of ablation was PV isolation; this was confirmed when Lasso mapping showed the disappearance of all PV potentials or the dissociation of PV potentials from LA activity.
  The ICM (Reveal XT, Medtronic Inc) was implanted the day of the ablation procedure or 1 week before.The Reveal XT was implanted in the parasternal area of the chest. The requirement for defining the exact final position was an R-wave amplitude ≥0.4 mV assessed through the Vector Check.

SUMMARY:
The aim of this study is to identify the most appropriate method for managing patients with AF recurrences after the first ablation procedure, through the diagnostic data stored by a subcutaneous AF monitor.

ELIGIBILITY:
Inclusion Criteria:

* highly symptomatic patients refractory to at least two antiarrhythmic drugs
* patients with sustained PAF episodes and/or history of PersAF interrupted with cardioversion.

Exclusion Criteria:

* congestive heart failure
* ejection fraction <35%
* left atrial diameter >60 mm
* previous ablation procedure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-02; Primary Completion 2010-02 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Freedom from atrial fibrillation or atrial flutter/tachycardia in Group 4 vs Group 3 | 12 months

SECONDARY OUTCOMES:
Freedom from AF in each group and the comparison of any group to each other | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny A Pokushalov, MD, PhD, Principal Investigator — State Research Institute of Circulation Pathology
Locations (1):
- State Research Institute of CIrculation Pathology, Novosibirsk, Russia

REFERENCES:
- [Result] Pokushalov E, Romanov A, Corbucci G, Artyomenko S, Turov A, Shirokova N, Karaskov A. Use of an implantable monitor to detect arrhythmia recurrences and select patients for early repeat catheter ablation for atrial fibrillation: a pilot study. Circ Arrhythm Electrophysiol. 2011 Dec;4(6):823-31. doi: 10.1161/CIRCEP.111.964809. Epub 2011 Sep 19. PMID 21930653